CLINICAL TRIAL: NCT04296006
Title: Neurobehavioral Mechanisms of Cocaine Choice
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Joshua A. Lile, Ph.D. (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor-Investigator, Joshua A. Lile, Ph.D., Professor of Behavioral Science, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: BED(In)(41); R01DA045023 (NIH)
Record Dates: First submitted 2020-03-02; First posted 2020-03-05 (Actual); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Cocaine Use Disorder
MeSH Terms: interventions — Cocaine

STUDY DESIGN:
Intervention Model Description: A placebo-controlled, randomized, within-subjects design will be used to assess cocaine-vs-money choice in cocaine use disordered subjects as a function of alternative reinforcer value.
Who Masked: Participant, Outcomes Assessor
Masking Description: Cocaine dose is administered under double-blind conditions. Available money value is not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- $0.25 alternative reinforcer value (Experimental): Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and an alternative monetary reinforcer are available during each trial. Each money value is tested in a separate session.
  Interventions: Behavioral: Money; Drug: Cocaine HCl
- $1.00 alternative reinforcer value (Experimental): Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and an alternative monetary reinforcer are available during each trial. Each money value is tested in a separate session.
  Interventions: Behavioral: Money; Drug: Cocaine HCl
- $4.00 alternative reinforcer value (Experimental): Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and an alternative monetary reinforcer are available during each trial. Each money value is tested in a separate session.
  Interventions: Behavioral: Money; Drug: Cocaine HCl

INTERVENTIONS:
Behavioral: Money — Three money values offered as alternatives to cocaine.
Drug: Cocaine HCl — 3 mg/70 kg is available as an alternative to money.

SUMMARY:
The objective of this protocol is to use a drug-vs-money choice task, reinforcement learning modeling and fMRI to determine the neurobehavioral and neurobiological decision-making "profile" associated with the decision to take cocaine and the reduced cocaine choice that occurs during a behavioral intervention (alternative money reinforcer) that models contingency management.

ELIGIBILITY:
Inclusion Criteria:

* Recent cocaine use, otherwise healthy

Exclusion Criteria:

* Laboratory results outside of clinically acceptable ranges, history of or current serious physical or psychiatric disease

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Lile, PhD, Principal Investigator — University of Kentucky
Locations (1):
- Laboratory of Human Behavioral Pharmacology, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects were lost to follow up and 4 subjects were screen fails. All 8 subjects who were admitted to the inpatient unit completed the three within-subjects experimental conditions.
Groups:
- The Impact of Alternative Reinforcer Magnitude on Cocaine vs Money Choice: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and varying amounts of money ($0.25, 1.00, 4.00) are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
Period: Overall Study
Arm/Group | The Impact of Alternative Reinforcer Magnitude on Cocaine vs Money Choice
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- The Effects of Alternative Reinforcer Magnitude on Cocaine vs Money Choice: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and varying amounts of money ($0.25, 1.00, 4.00) are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
Arm/Group | The Effects of Alternative Reinforcer Magnitude on Cocaine vs Money Choice
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 49 [44 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: The Number of Times Cocaine Was Selected in the Presence of a Monetary Reward Alternative
Description: The reinforcing effects of cocaine are determined using a reinforcement learning choice task. Subjects complete trials in which they could possibly receive the available cocaine dose or money. Reinforcing effects are measured for a fixed cocaine dose when three amounts of money are available as alternatives to cocaine. Each money value is tested in a separate session.
Time Frame: Choices occur across a 40 minute session
Population: People with cocaine use disorder
Measure: Mean (Standard Deviation); unit: number of choices
Groups:
- $0.25 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $0.25 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
- $1.00 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $1.00 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
- $4.00 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $4.00 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
Arm/Group | $0.25 Alternative Reinforcer Value | $1.00 Alternative Reinforcer Value | $4.00 Alternative Reinforcer Value
Number analyzed (Participants) | 8 | 8 | 8
number of choices | 110 (34) | 98 (17) | 90 (12)

ADVERSE EVENTS:
Time Frame: AEs were collected during the duration of data collection on three separate days.
Groups:
- $0.25 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $0.25 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
  This is a within-subjects study, but AE results are reported by each of the three experimental conditions (i.e., 3 separate alternative money conditions) that each subject completed on separate sessions.
- $1.00 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $1.00 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
  This is a within-subjects study, but AE results are reported by each of the three experimental conditions (i.e., 3 separate alternative money conditions) that each subject completed on separate sessions.
- $4.00 Alternative Reinforcer Value: Subjects complete 200 trials on a probabilistic concurrent choice procedure in which 3 mg/70 kg intravenous cocaine and $4.00 are available during each trial.
  Money: Three money values offered as alternatives to cocaine.
  Cocaine HCl: 3 mg/70 kg is available as an alternative to money.
  This is a within-subjects study, but AE results are reported by each of the three experimental conditions (i.e., 3 separate alternative money conditions) that each subject completed on separate sessions.
Arm/Group | $0.25 Alternative Reinforcer Value | $1.00 Alternative Reinforcer Value | $4.00 Alternative Reinforcer Value
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 1/8 | 1/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | $0.25 Alternative Reinforcer Value (N=8) | $1.00 Alternative Reinforcer Value (N=8) | $4.00 Alternative Reinforcer Value (N=8)
Elevated Heart Rate (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Elevated Blood Pressure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-02-11): https://cdn.clinicaltrials.gov/large-docs/06/NCT04296006/Prot_SAP_000.pdf